CLINICAL TRIAL: NCT03891784
Title: A Phase 2 Trial of the CDK4/6 Inhibitor Abemaciclib in Patients With Advanced and Refractory Well-Differentiated Gastroenteropancreatic Neuroendocrine Tumors (GEP NETs)
Brief Title: Abemaciclib in Treating Patients With Advanced, Refractory, and Unresectable Digestive System Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1004456; NCI-2019-01490 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9959 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced Digestive System Neuroendocrine Neoplasm; Digestive System Neuroendocrine Tumor; Foregut Neuroendocrine Tumor; Hindgut Neuroendocrine Tumor; Locally Advanced Unresectable Digestive System Neuroendocrine Neoplasm; Metastatic Digestive System Neuroendocrine Neoplasm; Midgut Neuroendocrine Tumor; Pancreatic Neuroendocrine Tumor; Refractory Digestive System Neuroendocrine Neoplasm
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Adenoma, Islet Cell | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (abemaciclib) (Experimental): Patients receive abemaciclib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: Verzenio; 1231929-97-7; 2-Pyrimidinamine

SUMMARY:
This phase II trial studies how well abemaciclib works in treating patients with digestive system neuroendocrine tumors that have spread to other places in the body, do not respond to treatment, and cannot be removed by surgery. Abemaciclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
Patients receive abemaciclib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 4 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed GEP NET, radiographically progressed on at least one line of standard therapy within the past 12 months

  * Primary tumors may be in: pancreas, foregut (esophagus, stomach, duodenum), midgut (small intestine, appendix), hindgut (large intestine, rectum), or unknown origin
  * Tumors may be functional (associated with clinical symptoms of hormone secretion) or non-functional
* Well-differentiated NET with low grade (Ki67 index < 3% or mitotic index < 2 mitoses/10 high power field [HPF]), intermediate grade (Ki67 index 3-20% or mitotic index 2-20 mitoses/10 HPF), or high grade (Ki67 21% to ≤ 55% of mitotic index 21-55% mitoses/10 HPF). In cases where pathology reports call out only a "high grade neuroendocrine carcinoma", such patients are eligible only if well differentiated status is confirmed by a board-certified pathologist AND Ki-67 is ≤ 55%
* Metastatic or locally advanced unresectable disease
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) as per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1
* Prior or concurrent therapy with somatostatin analogs (SSAs) is allowed. If concurrent therapy, dose must be stable for at least 2 months
* Patients with carcinoid syndrome must have symptoms controlled with stable doses of SSAs for at least 2 months

  * Telotristat is not allowed
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Able to swallow oral medications
* Absolute neutrophil count >= 1500/uL
* Platelet count >= 100,000/uL (without platelet transfusion for at least two weeks)
* Hemoglobin >= 8 g/dL (blood transfusion is not allowed the day before or on the day of study treatment)
* Total bilirubin =< 1.5 times upper limit of normal (ULN)
* Transaminases (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT]) =< 3 x upper limit of normal (ULN) (=< 5 x ULN if liver metastases)
* Patients with Gilbert's syndrome with a total bilirubin =< 2.0 times ULN and direct bilirubin within normal limits are permitted
* International normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x ULN
* Creatinine > 30 mL/min
* Ability to understand and sign the consent form
* Women of child-bearing potential must:

  * Have a negative serum pregnancy test within 7 days prior to initiation of treatment, and
  * Agree to use a highly effective method of contraception during the study and for at least 3 weeks following the last dose of study drug
* Men must be sterile or agree to use a highly effective method of contraception during the study and for at least 3 weeks following the last dose of study drug

Exclusion Criteria:

* Presence of poorly differentiated neuroendocrine carcinoma (NEC) or mixed adenoneuroendocrine carcinomas (MANECs)
* Prior treatment with abemaciclib or other CDK4/6 inhibitors
* Known hypersensitivity to abemaciclib or its components
* Receipt of any therapy or investigational agent within 4 weeks prior to study registration, except SSAs
* Any surgery, radiation, or embolization within 4 weeks
* Peptide receptor radionuclide therapy (PRRT) within 6 weeks
* Patients receiving other investigational agents
* Patients who have not recovered from adverse events of prior therapy to =< grade 1 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5), except for alopecia or grade =< 2 peripheral neuropathy prior to study treatment initiation. Subjects must have fully recovered from the acute effects of any prior radiotherapy
* Patients with untreated or symptomatic brain metastases (must be off corticosteroids for >= 4 weeks)
* Uncontrolled or untreated intercurrent illness including, but not limited to, active bacterial or fungal infection, congestive heart failure, severe/unstable angina, syncope of cardiac etiology, ventricular arrythmia (including but not limited to ventricular tachycardia, ventricular fibrillation), history of cardiac arrest, interstitial lung disease, severe dyspnea at rest or requiring oxygen supplementation, arterial or venous thrombotic event, pre-existing chronic condition resulting in baseline grade >= 2 diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures involving stomach or small bowel in the last 28 days, active peptic ulcer disease, Crohn's disease or ulcerative colitis
* Severe renal impairment (e.g. estimated creatinine clearance < 30ml/min)
* Known history of infection with human immunodeficiency virus (HIV)
* Active untreated infection with hepatitis B virus (i.e. hepatitis B surface antigen positive) or hepatitis C virus (i.e. hepatitis C antibody and ribonucleic acid [RNA] positive)
* Other malignancy diagnosed or recurrent in the past 3 years (except non-melanoma skin cancer and in-situ cervical cancer)
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 1 year after completion of study treatment
  ORR defined as complete or partial response as per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1, will be represented by a waterfall plot.

SECONDARY OUTCOMES:
Progression-free survival | From study registration to radiographic progression per RECIST v1.1 (investigator assessment), clinical progression, or death of any cause, assessed up to 1 year
  The distribution for survival times will be estimated using the method of Kaplan-Meier; associated landmark time percentages and the median value will be based on this. Confidence intervals for median values will use the Brookmeyer-Crowley method. Survival outcomes between carcinoid tumors and pancreatic neuroendocrine tumor (PNET)s will be compared using a log-rank test.
Overall survival | Time from study registration to death of any cause, assessed up to 1 year
  The distribution for survival times will be estimated using the method of Kaplan-Meier; associated landmark time percentages and the median value will be based on this. Confidence intervals for median values will use the Brookmeyer-Crowley method. Survival outcomes between carcinoid tumors and PNETs will be compared using a log-rank test.
Incidence of adverse events | Up to 30 days
  Safety will be evaluated by assessing the adverse events according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.

CONTACTS AND LOCATIONS:
Overall Officials: David B. Zhen, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - University of Colorado, Denver, Colorado
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT03891784/ICF_000.pdf